CLINICAL TRIAL: NCT03421535
Title: Sacroiliac Stretching Improves Glenohumeral Internal Rotational Deficit of the Opposite Shoulder in Baseball Players in a Randomized Control Study
Brief Title: Opposite SI Joint Stretching for GIRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Romano Orthopaedic Center (Other)
Responsible Party: Principal Investigator, Victor Romano, MD, Orthopaedic Surgeon, Romano Orthopaedic Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#2017-087
Record Dates: First submitted 2017-12-30; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Shoulder Impingement
Keywords: Glenohumeral internal rotational deficit; GIRD; Sleeper stretch; SI joint stretch
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: All 23 players of a minor league baseball team voluntarily participated in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each player was randomly assigned to either a sleeper stretch group or an opposite SI joint stretch group. The investigators were blinded to the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeper stretch group (Active Comparator): A certified athletic trainer supervised and observed the athlete as he performed the sleeper stretch on his dominant shoulder.
  Interventions: Procedure: Sleeper Stretch
- Opposite SI joint Stretch (Experimental): A certified athletic trainer supervised and observed the athlete as he performed the SI joint stretch opposite his dominant shoulder.
  Interventions: Procedure: Opposite SI joint Stretch

INTERVENTIONS:
Procedure: Sleeper Stretch — Internal Range of motion of dominant shoulder
  Arms: Sleeper stretch group
Procedure: Opposite SI joint Stretch — Internal range of motion of dominant shoulder
  Arms: Opposite SI joint Stretch

SUMMARY:
The purpose of this study is to investigate if stretching the contralateral sacroiliac (SI) joint improves GIRD in baseball players. Additionally, we aimed to compare our SI joint stretching regiment with a classically described sleeper stretch routine.

DETAILED DESCRIPTION:
Abstract:

Background:

Glenohumeral Internal Rotational Deficit (GIRD) is a well-documented finding in throwing athletes.

Hypothesis/Purpose:

The purpose of this study is to investigate if stretching the contralateral sacroiliac (SI) joint improves GIRD in baseball players. Additionally, the effect of the SI joint stretch will be compared to that of the classically described sleeper stretch.

Study Design:

Randomized Controlled Clinical Trial

Methods:

With the athlete supine and arm abducted 90o, internal rotation of both shoulders was measured in 23 minor league baseball players.

Next, each player randomly was assigned to either a control (sleeper stretch of dominant shoulder) or experimental (stretch of the SI joint contralateral to the dominant shoulder) group supervised by a certified athletic trainer. The players performed their own stretches.

Finally, the initial two investigators, unaware of to which group the player was assigned, re-measured the end-range internal rotation of each athlete's dominant shoulder.

ELIGIBILITY:
Inclusion Criteria:

* All members a minor league baseball team

Exclusion Criteria:

* Any active shoulder or back injury or history of shoulder or back injury

Ages: 23 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Shoulder internal ROM after stretching opposite SI joint | Measurement made within 30 minutes of stretching
  Internal range of motion of dominant shoulder after stretching opposite SI joint

SECONDARY OUTCOMES:
Shoulder Internal ROM after sleeper stretch | Measurement made with 30 minutes of stretching
  Internal range of motion of dominant shoulder after sleeper stretch

CONTACTS AND LOCATIONS:
Overall Officials: Victor Romano, Principal Investigator — Romano Orthopaedic Center
Locations (1):
- Romano Orthopaedic Center, Oak Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Bigliani LU, Codd TP, Connor PM, Levine WN, Littlefield MA, Hershon SJ. Shoulder motion and laxity in the professional baseball player. Am J Sports Med. 1997 Sep-Oct;25(5):609-13. doi: 10.1177/036354659702500504. PMID 9302464